CLINICAL TRIAL: NCT03968016
Title: Reference Interval Validation of High-Sensitivity Cardiac Troponin T Assay in Thai Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Troponin T
Record Dates: First submitted 2019-05-09; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Diagnoses Disease
Keywords: Acute Myocardial Infarction; Cardiac marker; Troponin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Placebo Comparator): Control group
  Interventions: Device: SYSMEX HLSCL
- Stable heart disease (Active Comparator): Stable heart disease and non-hospitalized
  Interventions: Device: SYSMEX HLSCL

INTERVENTIONS:
Device: SYSMEX HLSCL — Diagnostic device

SUMMARY:
The investigators aimed to study the cut-off of high sensitivity troponin T using SYSMEX HLSCL Machine in Thai population at percentile 99.

ELIGIBILITY:
For healthy group

Inclusion Criteria:

* Group 1: Aged 18 - 40 years
* Group 2: Aged > 40 - 70 years
* A presumably healthy population will define from a health questionnaire

Exclusion Criteria:

* Heart diseases
* Renal diseases (CKD or recent AKI)
* History of pulmonary embolism

For Patient group with stable heart diseases

Inclusion Criteria:

* Aged > 40 - 70 years
* Stable heart disease individuals will be evaluated by cardiologist
* Non hospitalized (OPD settings)

Exclusion Criteria:

* Stable heart diseases with ACS
* Renal diseases (CKD or recent AKI)
* History of pulmonary embolism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Measurement of high sensitivity-troponin T level | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand